CLINICAL TRIAL: NCT05666388
Title: Rescue Stenting in the Severe Atherosclerotic Stenosis After the Failure of Intravenous Thrombolysis: an Initial Vietnamese Report
Brief Title: Rescue Stenting in the Severe Atherosclerotic Stenosis After the Failure of Intravenous Thrombolysis
Acronym: RESFIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Can Tho Stroke International Services Hospital (Other)
Responsible Party: Principal Investigator, Dr. Cuong Tran Chi, Director - Doctor, Can Tho Stroke International Services Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RESFIT study
Record Dates: First submitted 2022-12-17; First posted 2022-12-27 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Ischemic Stroke, Acute; Stent Stenosis; Thrombosis
Keywords: Ischemic stroke; Rescue stenting; Intravenous thrombolysis; Dual antiplatelet therapy
MeSH Terms: conditions — Ischemic Stroke; Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rescue stenting (RESFIT) (Experimental): Rescue stenting in the severe atherosclerotic stenosis after the failure of intravenous thrombolysis (RESFIT)
  Interventions: Procedure: Rescue stenting

INTERVENTIONS:
Procedure: Rescue stenting — Rescue stenting in the severe atherosclerotic stenosis after the failure of intravenous thrombolysis (RES

SUMMARY:
Intravenous (IV) recombinant tissue plasminogen activator is the standard of care for patients with acute ischemic stroke (AIS) who present to the hospital within 4.5 hours of symptom onset. However, IV thrombolysis, even bridging thrombolysis (combining intravenous thrombolysis and mechanical thrombectomy) has limited efficacy among patients who had occlusive lesions associated with highgrade arterial stenosis requiring revascularization to improve neurological deficits. The investigators evaluated whether rescue stenting results in good outcomes among patients after the failure of intravenous thrombolysis and bridging thrombolysis.

DETAILED DESCRIPTION:
Stroke is the second most common cause of death worldwide, with an annual mortality rate of approximately 5.5 million. Depending on the timing of presentation, intravenous (IV) administration of recombinant tissue plasminogen activator can be an effective treatment, but is most effective when used between 3 and 4.5 hours of symptom onset. Bridging thrombolysis, which describes the combination of IV thrombolysis and mechanical thrombectomy, can lead to long-term functional independence after 90 days with higher recanalization success rates than IV thrombolysis alone without increased risk. The HERMES meta-analysis of fve trials (MR CLEAN, ESCAPE, REVASCAT, SWIFT PRIME, and EXTEND IA) indicated the potential benefits of mechanical thrombectomy (MT) in case of proximal circulation occlusions. The recanalization failure rate of this treatment, defined as a modified Thrombolysis in Cerebral Ischemia (mTICI) score of 2a or worse, remained high, ranging from 13% to 29%, and most patients experienced poor clinical outcomes. Permanent stent placement has been suggested as a potential approach for achieving successful recanalization, which is the goal of endovascular therapy in the early management of acute ischemic stroke (AIS). However, the risk of intracranial hemorrhage associated with the combined use of IV thrombolysis and a loading dose of dual antiplatelet therapy (DAPT) increases when rescue stenting is applied. The investigators hypothesize that stent deployment might serve as a feasible treatment for large artery occlusion after the failure of intravenous thrombolysis and bridging thrombolysis.

ELIGIBILITY:
Inclusion Criteria:

* Acute ischemic stroke who underwent rescue stenting for large vessel occlusions underlying severe atherosclerotic stenosis after the failure of intravenous alteplase therapy.
* Absence of intracranial hemorrhage.

Exclusion Criteria:

* Premorbid modified Rankin Scale (mRS) ≥ 2
* Initiation to rescue stenting beyond 24 hours after symptom onset

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
The incidence of hemorrhagic transformation | 24 hours after rescue intracranial stenting.
  Hemorrhagic transformation was accessed by CT scan or MRI.
The rate of good outcomes at 3-month follow-up | 3 months
  The good 3-month outcome rate was accessed by modified Rankin Score (mRS) < 3.

CONTACTS AND LOCATIONS:
Overall Officials: Cuong C Tran, Doctor, Study Chair — Can Tho Stroke International Services General Hospital
Locations (1):
- Can Tho SIS Hospital, Can Tho, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tran CC, Le MT, Baxter BW, Nguyen-Luu G, Ngo MT, Nguyen-Dao NH, Duong-Hoang L, Mai-Van M, Nguyen MD. Rescue intracranial stenting in acute ischemic stroke: a preliminary Vietnamese study. Eur Rev Med Pharmacol Sci. 2022 Oct;26(19):6944-6952. doi: 10.26355/eurrev_202210_29875. PMID 36263574
- [Background] Sallustio F, Koch G, Rocco A, Rossi C, Pampana E, Gandini R, Meschini A, Diomedi M, Stanzione P, Di Legge S. Safety of early carotid artery stenting after systemic thrombolysis: a single center experience. Stroke Res Treat. 2012;2012:904575. doi: 10.1155/2012/904575. Epub 2011 Aug 8. PMID 21860810
- [Background] Kwon DH, Jang SH, Park H, Sohn SI, Hong JH. Emergency Cervical Carotid Artery Stenting After Intravenous Thrombolysis in Patients With Hyperacute Ischemic Stroke. J Korean Med Sci. 2022 May 16;37(19):e156. doi: 10.3346/jkms.2022.37.e156. PMID 35578588
- [Background] Stracke CP, Fiehler J, Meyer L, Thomalla G, Krause LU, Lowens S, Rothaupt J, Kim BM, Heo JH, Yeo LLL, Andersson T, Kabbasch C, Dorn F, Chapot R, Hanning U. Emergency Intracranial Stenting in Acute Stroke: Predictors for Poor Outcome and for Complications. J Am Heart Assoc. 2020 Mar 3;9(5):e012795. doi: 10.1161/JAHA.119.012795. Epub 2020 Mar 3. PMID 32122218